CLINICAL TRIAL: NCT02649933
Title: Detection of Sleep Apnea Syndrome (OSA) With Watch PAT 200 in Pregnant Women and Assessment of Impact of OSA on Intra-uterine Fetal Growth and Maternal Well-being
Brief Title: Detection of Sleep Apnea Syndrome (OSA) in Pregnant Women and Assessment of Impact of OSA on Pregnancy Course
Status: Terminated | Type: Observational
Why Stopped: one investigator left the study site
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Marie Bruyneel, chef de clinique service de pneumologie, Centre Hospitalier Universitaire Saint Pierre
Other Study IDs: AK/14-11-105/4434
Record Dates: First submitted 2015-12-17; First posted 2016-01-08 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Pregnancy; Sleep Apnea Syndrome; Obstructive Sleep Apnea
Keywords: pregnancy; obstructive sleep apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Watch PAt 200: obese pregnant women, pregnancy between 12 and 15 weeks
  Interventions: Device: Watch PAT 200

INTERVENTIONS:
Device: Watch PAT 200 — screening of OSA with Watch PAT 200

SUMMARY:
To assess prevalence of obstructive sleep apnea during pregnancy and its impact on prgnancy course and materno foetal wellbeing.

DETAILED DESCRIPTION:
During pregnancy, obstructive sleep apnea (OSA) prevalence is estimated between 5% and 15% and is associated with maternal and fetal comorbidities such as preeclampsia, neonatal intensive care admission , fetal growth retardation , preterm birth but even if growing, literature is still relatively poor about this topic.

To date, there is no systematic screening of OSA performed in at-risk pregnant women (obesity, hypertension, diabetes, fetal growth retardation, suggestive symptoms), probably mainly because of polysomnography complexity and accessibility.

As in non pregnant woman, OSA must be treated adequately during pregnancy. Continuous positive airway pressure (CPAP) is the reference treatment for severe OSA. This device, by blowing air under pressure in upper airways, via a nasal of an oro-nasal mask, is able to alleviate the upper airway collapse responsible for the occurrence of obstructive sleep apnea. It has been proven to offer a survival benefit in patients with severe disease and to improve sleep quality, cardiovascular variables and health-related quality of life . CPAP have been shown to improve fetal well-being in pre-eclampsia .

Oral appliance can be an alternative for mild to moderate disease and in patients who do not tolerate CPAP. Positional counselling can be sufficient in case of mild to moderate positional OSA. Associated behavioural strategies (diet and exercise) are always recommended in case of excessive weight. Surgical treatments are dedicated to patients with specific anatomic problems but cannot be performed during pregancy.

Aim of the study:

The primary aim of this study is to screen OSA in at risk pregnant women with Watch-PAT 200, a simplified sleep study tool used on ambulatory mode and able to detect accurately OSA in suspected patients. As secondary aim, we will observe the impact of OSA on a composite endpoint assessing materno-fetal wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* 12-15weeks of pregnancy
* obese (body mass index>30)

Exclusion Criteria:

* known sleep apnea syndrome
* mental illness, deficiency

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: pregnant women, 12-15weeks of pregnancy, obese (body mass index>30)
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2015-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
prevalence of sleep apnea syndrome (OSA) in obese pregnant women | 1 month
  Positive OSA on Watch Pat 200 must be confirmed by polysomnography

SECONDARY OUTCOMES:
composite score assessing pregnancy course and materno-foetal complications | 6 months
  assessment of one composite score componed by on several parameters including Apgar Score,fœtal anoxia, intra-uterine growth retardation, low birth weight, prematurity, placental abruption,preeclamspia, foetal death In Utero

CONTACTS AND LOCATIONS:
Locations (1):
- CHU St Pierre, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No